CLINICAL TRIAL: NCT01629511
Title: Clofarabine, Gemcitabine, and Busulfan Followed by Allogeneic Stem Cell Transplantation for Chronic Lymphocytic Leukemia (CLL)
Brief Title: Allogeneic Stem Cell Transplant for CLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0249; NCI-2018-01798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0249 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Richter Syndrome
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Clofarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Gemcitabine; Methotrexate; merphos; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (combination chemotherapy, stem cell transplant) (Experimental): Participants receive gemcitabine IV over 10-25 minutes on days -6 and -4, clofarabine IV over 1 hour and busulfan IV over 3 hours on days -6 to -3. Participants with matched unrelated donors also receive anti-thymocyte globulin IV over 4 hours on days -3 to -1. Starting day -2, participants receive tacrolimus PO daily for up to 6 months. Participants undergo hematopoietic allogeneic stem cell transplant on day 0, then receive methotrexate IV over 15 minutes on days 1, 3, 6 and 11, and filgrastim SC QD beginning 1 week after transplant until blood cell levels return to normal.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Clofarabine; Biological: Filgrastim; Drug: Gemcitabine; Drug: Methotrexate; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo stem cell transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Tacrolimus — Given PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase I/II trial studies the best dose and side effects of gemcitabine and how well it works with clofarabine and busulfan and donor stem cell transplant in treating participants with chronic lymphocytic leukemia. Drugs used in chemotherapy, such as gemcitabine, clofarabine, and busulfan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of gemcitabine when administered with busulfan and clofarabine.

II. To estimate the day 100 treatment-related mortality (TRM) for the preparative regimen busulfan, clofarabine, and gemcitabine followed by allogeneic hematopoietic cell transplantation (HCT) for patients with chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. To determine the rate of progression-free survival (PFS), graft versus host disease (GVHD), engraftment, and overall survival (OS) for this treatment regimen at one year post treatment completion.

OUTLINE: This is a dose-escalation study of gemcitabine.

Participants receive gemcitabine intravenously (IV) over 10-25 minutes on days -6 and -4, clofarabine IV over 1 hour and busulfan IV over 3 hours on days -6 to -3. Participants with matched unrelated donors also receive anti-thymocyte globulin IV over 4 hours on days -3 to -1. Starting day -2, participants receive tacrolimus orally (PO) daily for up to 6 months. Participants undergo hematopoietic allogeneic stem cell transplant on day 0, then receive methotrexate IV over 15 minutes on days 1, 3, 6 and 11, and filgrastim subcutaneously (SC) once daily (QD) beginning 1 week after transplant until blood cell levels return to normal.

After completion of study treatment, participants are followed up at 3, 6 and 12 months, then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic leukemia, prolymphocytic leukemia, or Richter's transformation who are eligible for allogeneic transplantation and are not eligible for protocols of higher priority
* A 10/10 HLA matched (high resolution typing at A, B, C, DRB1, DQ1) sibling or unrelated donor
* Left ventricular ejection fraction (EF) > 40%
* Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and corrected diffusion capacity of the lung for carbon monoxide (DLCO) > 40%
* Serum creatinine < 1.6 mg/dL
* Serum bilirubin < 2 X upper limit of normal
* serum glutamate pyruvate transaminase (SGPT) < 2X upper limit of normal
* Voluntary signed, written Institutional Review Board (IRB)-approved informed consent
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Patient with active central nervous system (CNS) disease
* Pregnant (positive beta human chorionic gonadotropin [HCG] test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Known infection with human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV)-I, hepatitis B, or hepatitis C
* Active uncontrolled bacterial, viral or fungal infections
* Patient has received other investigational drugs within 1 week before enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Hosing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at MD Anderson clinic starting on November 21, 2012 on Phase I of the study. No participants were enrolled on Phase II.
Groups:
- Gemcitabine Dose Level 1: Gemcitabine 100 mg/m2 IV preceded by loading dose of 75 mg/m2 for 2 days + Busulfan(adjusted Pharmacokinetic dosing) IV for 4 days + Clofarabine 30 mg/m2 IV for 4 days + Thymoglobulin 4mg/kg(Matched Unrelated Donor patients only) IV for 3 days + Stem Cell Transplant
- Gemcitabine Dose Level 2: Gemcitabine 150 mg/m2 IV preceded by loading dose of 75 mg/m2 for 2 days + Busulfan(adjusted Pharmacokinetic dosing) IV for 4 days + Clofarabine 30 mg/m2 IV for 4 days + Thymoglobulin 4mg/kg(Matched Unrelated Donor patients only) IV for 3 days + Stem Cell Transplant
- Gemcitabine Dose Level 3: Gemcitabine 200 mg/m2 IV preceded by loading dose of 75 mg/m2 for 2 days + Busulfan(adjusted Pharmacokinetic dosing) IV for 4 days + Clofarabine 30 mg/m2 IV for 4 days + Thymoglobulin 4mg/kg(Matched Unrelated Donor patients only) IV for 3 days + Stem Cell Transplant
- Gemcitabine Dose Level 4: Gemcitabine 250 mg/m2 IV preceded by loading dose of 75 mg/m2 for 2 days + Busulfan(adjusted Pharmacokinetic dosing) IV for 4 days + Clofarabine 30 mg/m2 IV for 4 days + Thymoglobulin 4mg/kg(Matched Unrelated Donor patients only) IV for 3 days + Stem Cell Transplant
Period: Overall Study
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Started | 4 | 0 | 8 | 3
Completed | 4 | 0 | 8 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients age 18-70 with CLL, PLL, or Richter's Transformation who were eligible for allogeneic transplantation
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4 | Total
Number analyzed (Participants) | 4 | 0 | 8 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 7 | 3 | 13
  >=65 years | 1 | 0 | 1 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 67] |  | 57.5 [36 to 67] | 60 [59 to 61] | 59 [39 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 0 | 5
  Male | 1 | 0 | 6 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 2 | 2 | 5
  Unknown or Not Reported | 3 | 0 | 6 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 0 | 8 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 0 | 8 | 3 | 15
Disease Category [Count of Participants; unit: Participants]
  Diseases : Chronic Lymphocytic Leukemia (CLL) | 3 | 0 | 5 | 1 | 9
  Diseases : Prolymphocytic Leukemia (PLL) | 1 | 0 | 2 | 2 | 5
  Diseases: Richter's | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 100 Day Treatment Related Mortality (TRM)
Description: Number of deaths related to treatment by day 100 post allogeneic transplant
Time Frame: 100 days post transplant
Population: No participants were treated at dose level 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 4 | 0 | 8 | 3
Participants
  Infection | 0 | 0 | 0 | 0
  Graft versus Host Disease (GVHD) | 0 | 0 | 1 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: To find the maximum tolerated dose (MTD) of Gemcitabine when administered with Busulfan & Clofarabine
Time Frame: Enrollment up to day 30 post transplant
Population: MTD analysis was for Phase II. Data were not collected.
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Will be estimated by the method of Kaplan and Meier. Time-to-event distributions as function of patient baseline covariates will be evaluated using Bayesian time-to-event regression modeling.
Time Frame: Up to 1 year post transplant
Population: All participants were registered on Phase I.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 4 | 0 | 8 | 3
Participants | 3 | 0 | 4 | 2

4. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: Number of patients without any relapse post treatment completion
Time Frame: Up to 1 year post transplant
Population: Analysis was for Phase II. No analysis was done due to low accrual on Phase I.
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Time-to-engraftment
Description: The number of days until participants by dose level reach engraftment.
Time Frame: 30 days post transplant
Population: No participants were treated at dose level 2.
Measure: Number; unit: participants
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 4 | 0 | 8 | 3
participants
  Day 10 | 1 |  | 2 | 0
  Day 11 | 2 |  | 4 | 0
  Day 12 | 1 |  | 0 | 1
  Day 13 | 0 |  | 1 | 0
  Day 15 | 0 |  | 0 | 1
  Day 17 | 0 |  | 0 | 1
  <10 days - Graft Failure | 0 |  | 1 | 0

6. Other Pre Specified Outcome: Acute and Chronic Graft Verse Host Disease (GvHD)
Description: GvHD (Graft versus Host Disease) occurs when immune cells transplanted from a non-identical donor (graft) recognizes the transplant recipient (the host) as foreign, thereby initiating an immune reaction in the transplant recipient. Acute GvHD typically occurs around the time of engraftment and manifests in skin, GI system, and liver abnormalities. Chronic GvHD is defined by manifestations such as ocular, oral, lung, sclerosis skin, failure to thrive, fascia, cholestasis in liver, esophagus strictures.
Time Frame: Up to 1 year post transplant
Population: Analysis was for Phase II. No analysis was done due to low accrual on Phase I.
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 100 Days post transplant
Description: At Gemcitabine Dose Level 2, there were no participants at that dose level and so the number of participants at risk for adverse events is zero.
Arm/Group | Gemcitabine Dose Level 1 | Gemcitabine Dose Level 2 | Gemcitabine Dose Level 3 | Gemcitabine Dose Level 4
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/0 | 1/8 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 8/8 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Dose Level 1 (N=4) | Gemcitabine Dose Level 2 (N=0) | Gemcitabine Dose Level 3 (N=8) | Gemcitabine Dose Level 4 (N=3)
Hypertension (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Fluid Overload (General disorders) | 4 (4) | 0 (0) | 5 (5) | 3 (3)
Fever (General disorders) | 4 (5) | 0 (0) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Mucositis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (8) | 3 (3)
Elevated Creatinine (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 3 (5) | 0 (0) | 6 (6) | 3 (4)
Elevated Bilirubin (Hepatobiliary disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Infection (Infections and infestations) | 4 (8) | 0 (0) | 8 (15) | 3 (7)
Neutropenic Fever (General disorders) | 3 (3) | 0 (0) | 7 (7) | 2 (2)
Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Acute Graft versus Host Disease (General disorders) | 3 (5) | 0 (0) | 3 (7) | 2 (5)
Chronic Graft versus Host Disease (General disorders) | 2 (3) | 0 (0) | 3 (8) | 2 (8)
Secondary Graft Failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Primary Graft Failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed. This study never moved to Phase II, therefore was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT01629511/Prot_SAP_000.pdf